CLINICAL TRIAL: NCT02828124
Title: A Phase 1/2 Study of BMS-986183 in Subjects With Advanced Hepatocellular Carcinoma
Brief Title: A Study of the Safety and Tolerability of BMS-986183 in Patients With Liver Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA015-003
Record Dates: First submitted 2016-07-07; First posted 2016-07-11 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation Monotherapy (Experimental)
  Interventions: Biological: BMS-986183
- Dose Expansion Monotherapy (Experimental)
  Interventions: Biological: BMS-986183
- Dose Escalation Combination Therapy (Experimental)
  Interventions: Biological: BMS-986183; Biological: Nivolumab
- Dose Expansion Combination Therapy (Experimental)
  Interventions: Biological: BMS-986183; Biological: Nivolumab

INTERVENTIONS:
Biological: BMS-986183 — specified dose on specified days
Biological: Nivolumab — specified dose on specified days
  Other Names: BMS-936558; Opdivo
  Arms: Dose Escalation Combination Therapy; Dose Expansion Combination Therapy

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of BMS-986183 in patients with liver cancer.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Must have advanced liver cancer that cannot be treated with surgery or other local methods
* Liver cancer is confirmed by a microscopic examination of tissue
* Liver disease is classified as 'A' by a standard method called Child-Pugh score
* Daily living abilities are classified as '0 or 1' by a standard method from the Eastern Cooperative Oncology Group (ECOG)
* Women must use contraception

Exclusion Criteria:

* Prior liver transplant
* Increase in blood pressure in some of the veins entering the liver
* Cancer that has spread to the brain or the layers of tissue that cover the brain or spinal cord
* Infection with both hepatitis B and C, both hepatitis D and B, infection with HIV, or other infections
* Disease of the heart or blood vessels around the heart
* Active cancers within the last 2 years
* No more than 2 prior systemic treatments or other investigational agents except PD-1/PD-L1 or Ipilimumab (Part 2)
* Currently on anti-platelet or anti-coagulation therapy
* Radiotherapy within 4 weeks of treatment
* Any major allergies

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Local Institution, Ottawa, Ontario, Canada
- Local Institution, Singapore, Singapore
- Local Institution, Seoul, South Korea
- Local Institution, Taipei, Taiwan

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 10 subjects were treated in this study. All 10 subjects were enrolled in BMS-986183 escalation (Part 1)
Groups:
- BMS-986183 3 mg; BMS-986183 9 mg; BMS-986183 18 mg; BMS-986183 36 mg: Dose escalation in combination with Nivolumab
Period: Overall Study
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Started | 1 | 2 | 1 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 1 | 6
Not completed — Disease Progression | 1 | 2 | 1 | 4
Not completed — AE Unrelated to Study Drug | 0 | 0 | 0 | 1
Not completed — Subject Withdrew Consent | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All treated paritcipants
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg | Total
Number analyzed (Participants) | 1 | 2 | 1 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All treated participants
  Years | 56.0 (NA) — Insufficient number of participants with events | 67.5 (4.9) | 57.0 (NA) — Insufficient number of participants with events | 49.5 (8.6) | 54.5 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    Female | 0 | 0 | 0 | 1 | 1
    Male | 1 | 2 | 1 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    White | 0 | 0 | 0 | 1 | 1
    Black or African American | 0 | 0 | 0 | 0 | 0
    Asian | 1 | 2 | 1 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events at Its Worst Grade
Description: Evaluated by comparing the incidence of Adverse Events (AEs) among subjects using their assigned treatment for at least one day.
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Incidence of Serious Adverse Events at Its Worst Grade
Description: Evaluated by comparing the incidence of Serious Adverse Events (SAEs) among subjects using their assigned treatment for at least one day.
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Primary Outcome: Incidence of Adverse Events Leading to Discontinuation
Description: Evaluated by comparing the incidence of Adverse Events leading to discontinuation among subjects using their assigned treatment for at least one day.
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Primary Outcome: Incidence of Adverse Events Leading to Death
Description: Evaluated by comparing the incidence of Adverse Events leading to death among subjects using their assigned treatment for at least one day.
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Primary Outcome: Incidence of Laboratory Test Toxicity Grade Shifting From Baseline
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Best Overall Response (BOR)
Description: Defined as BOR designation over the study as a whole, recorded between the dates of first dose until the last tumor assessment prior to subsequent therapy. CR or PR determinations included in the BOR assessment must be confirmed by a second scan performed no less than 4 weeks after the criteria for response are first met.
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Overall Response Rate (ORR)
Description: Defined as the total number of subjects whose BOR is either a CR or PR divided by the total number of subjects in the population of interest
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Duration of Response (DoR)
Description: Defined as the time between the date of first response and the subsequent date of objectively documented disease progression or death, whichever occurs first. For those subjects who remain alive and have not progressed or received subsequent therapy, DoR will be censored on the date of last tumor assessment
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Progression Free Survival (PFS)
Description: Defined as the time from the first dose of study drug to the date of the first objective documentation of tumor progression or death due to any cause. Subjects who did not progress nor died will be censored on the date of their last tumor assessment. Subjects who did not have any on-study tumor assessments will be censored on the date of the first dose of study drug.
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: PFS Rate at Week 't'
Description: Defined as the proportion of subjects who remain progression free and surviving at 't' weeks (t=12, 24, 36, etc). The proportion will be calculated by the product-limit method (Kaplan-Meier [K-M] estimate) which takes into account censored data
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Maximum Observed Concentration (Cmax)
Description: To characterize the PK of the total antibody [unconjugated antibody + antibody conjugated to tubulysin or antibody conjugated to any tubulysin metabolites], active ADC [antibody conjugated to tubulysin], and unconjugated tubulysin) of BMS-986183 as monotherapy and in combination with nivolumab will be measured by Cmax
Time Frame: From first does up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Time of Maximum Observed Concentration (Tmax)
Description: to characterize the PK of the total antibody [unconjugated antibody + antibody conjugated to tubulysin or antibody conjugated to any tubulysin metabolites], active ADC [antibody conjugated to tubulysin], and unconjugated tubulysin) of BMS-986183 as monotherapy and in combination with nivolumab will be measured by Tmax.
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to T of the Last Quantifiable Concentration [AUC(0-T)]
Description: to characterize the PK of the total antibody [unconjugated antibody + antibody conjugated to tubulysin or antibody conjugated to any tubulysin metabolites], active ADC [antibody conjugated to tubulysin], and unconjugated tubulysin) of BMS-986183 as monotherapy and in combination with nivolumab will be measured by AUC(0-T)]
Time Frame: First does up to appromimately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Area Under the Concentration-time Curve in 1 Dosing Interval [AUC(TAU)]
Description: To characterize the PK of the total antibody [unconjugated antibody + antibody conjugated to tubulysin or antibody conjugated to any tubulysin metabolites], active ADC [antibody conjugated to tubulysin], and unconjugated tubulysin) of BMS-986183 as monotherapy and in combination with nivolumab will be measured by AUC(TAU).
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Concentration at the End of a Dosing Interval (Ctau)
Description: To characterize the PK of the total antibody [unconjugated antibody + antibody conjugated to tubulysin or antibody conjugated to any tubulysin metabolites], active ADC [antibody conjugated to tubulysin], and unconjugated tubulysin) of BMS-986183 as monotherapy and in combination with nivolumab will be measured by
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Trough Observed Concentration, Including Predose Concentrations and Ctau (Ctrough)
Description: to characterize the PK of the total antibody [unconjugated antibody + antibody conjugated to tubulysin or antibody conjugated to any tubulysin metabolites], active ADC [antibody conjugated to tubulysin], and unconjugated tubulysin) of BMS-986183 as monotherapy and in combination with nivolumab will be measured by (Ctrough)
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Total Body Clearance (CLT)
Description: to characterize the PK of the total antibody [unconjugated antibody + antibody conjugated to tubulysin or antibody conjugated to any tubulysin metabolites], active ADC [antibody conjugated to tubulysin], and unconjugated tubulysin) of BMS-986183 as monotherapy and in combination with nivolumab will be measured by CLT
Time Frame: First dose to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Apparent Volume of Distribution at Steady-state (Vss)
Description: to characterize the PK of the total antibody [unconjugated antibody + antibody conjugated to tubulysin or antibody conjugated to any tubulysin metabolites], active ADC [antibody conjugated to tubulysin], and unconjugated tubulysin) of BMS-986183 as monotherapy and in combination with nivolumab will be measured by Vss
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

19. Secondary Outcome: Volume of Distribution of Terminal Phase (Vz)
Description: (to characterize the PK of the total antibody [unconjugated antibody + antibody conjugated to tubulysin or antibody conjugated to any tubulysin metabolites], active ADC [antibody conjugated to tubulysin], and unconjugated tubulysin) of BMS-986183 as monotherapy and in combination with nivolumab will be measured by Vz.
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

20. Secondary Outcome: Accumulation Index; Ratio of Cmax at Steady-state to Cmax After the First Dose (AI_Cmax)
Description: to characterize the PK of the total antibody [unconjugated antibody + antibody conjugated to tubulysin or antibody conjugated to any tubulysin metabolites], active ADC [antibody conjugated to tubulysin], and unconjugated tubulysin) of BMS-986183 as monotherapy and in combination with nivolumab will be measured by AI_Cmax.
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

21. Secondary Outcome: Accumulation Index; Ratio of Ctau at Steady-state to Ctau After the First Dose (AI_Ctau)
Description: to characterize the PK of the total antibody [unconjugated antibody + antibody conjugated to tubulysin or antibody conjugated to any tubulysin metabolites], active ADC [antibody conjugated to tubulysin], and unconjugated tubulysin) of BMS-986183 as monotherapy and in combination with nivolumab will be measured by AI_Ctau.
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

22. Secondary Outcome: Accumulation Index; Ratio of AUC(TAU) at Steady-state to AUC(TAU) After the First Dose [AI_AUC(TAU)]
Description: To characterize the PK of the total antibody [unconjugated antibody + antibody conjugated to tubulysin or antibody conjugated to any tubulysin metabolites], active ADC [antibody conjugated to tubulysin], and unconjugated tubulysin) of BMS-986183 as monotherapy and in combination with nivolumab will be measured by AI_AUC(TAU).
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

23. Secondary Outcome: Average Concentration Over a Dosing Interval Calculated by Dividing AUC(TAU) at Steady State by Tau (Css,Ave)
Description: To characterize the PK of the total antibody [unconjugated antibody + antibody conjugated to tubulysin or antibody conjugated to any tubulysin metabolites], active ADC [antibody conjugated to tubulysin], and unconjugated tubulysin) of BMS-986183 as monotherapy and in combination with nivolumab will be measured by Css,avg.
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

24. Secondary Outcome: Terminal Half-life (T-HALF)
Description: to characterize the PK of the total antibody [unconjugated antibody + antibody conjugated to tubulysin or antibody conjugated to any tubulysin metabolites], active ADC [antibody conjugated to tubulysin], and unconjugated tubulysin) of BMS-986183 as monotherapy and in combination with nivolumab will be measured by T-HALF.
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

25. Secondary Outcome: Changes in QTcF (ΔQTcF) From Baseline
Description: To assess the effect of dosage regimen and exposure [active ADC and unconjugated tubulysin] of BMS-986183 as monotherapy on the QT interval.
Time Frame: Baseline up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

26. Secondary Outcome: Incidence of Positive Anti-drug Antibody (ADA)
Description: The immunogenicity of BMS-986183 (as monotherapy and in combination with nivolumab) will be measured by assessment of the presence or absence of specific ADA to BMS-986183. The incidence of positive ADA will be calculated.
Time Frame: First dose up to approximately 24 months
Population: The study was terminated and data is not reported for privacy reasons.
Arm/Group | BMS-986183 3 mg | BMS-986183 9 mg | BMS-986183 18 mg | BMS-986183 36 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose up to approximately 24 months
Groups:
- BMS-986183 ESC 3 mg; BMS-986183 ESC 9 mg; BMS-986183 ESC 18 mg; BMS-986183 ESC 36 mg: Dose escalation in combination with Nivolumab
Arm/Group | BMS-986183 ESC 3 mg | BMS-986183 ESC 9 mg | BMS-986183 ESC 18 mg | BMS-986183 ESC 36 mg
All-Cause Mortality (participants affected / at risk) | 0/1 | 2/2 | 0/1 | 5/6
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2 | 1/1 | 2/6
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 1/1 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986183 ESC 3 mg (N=1) | BMS-986183 ESC 9 mg (N=2) | BMS-986183 ESC 18 mg (N=1) | BMS-986183 ESC 36 mg (N=6)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986183 ESC 3 mg (N=1) | BMS-986183 ESC 9 mg (N=2) | BMS-986183 ESC 18 mg (N=1) | BMS-986183 ESC 36 mg (N=6)
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 1 | 1 | 1 | 3
Pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (2):
  • Study Protocol (2017-05-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT02828124/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT02828124/SAP_001.pdf